CLINICAL TRIAL: NCT01593709
Title: Screening of Volunteers for Clinical Trials of Investigational and Licensed Vaccines, Antiviral Products, or Live Virus Challenge Studies
Brief Title: Volunteer Screening for Vaccine and Antivirals Clinical Trials
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 120121; 12-I-0121
Record Dates: First submitted 2012-05-05; First posted 2012-05-08 (Estimated); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Normal Physiology
Keywords: Anti-infective agents; ANTI-VIRAL AGENTS; Healthy Volunteers

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort 1: Healthy adults; age 18 or older

SUMMARY:
Background:

- Vaccines and antiviral therapies are critical for preventing and treating viral diseases. Testing these vaccines and drugs often requires healthy volunteers. To ensure that volunteers are healthy and eligible to participate in these studies, they will be screened before the start of the study. This screening may involve a medical history, physical exam, and blood test. Other samples may also be collected. This study will help identify volunteers who are eligible to participate in vaccine or antiviral therapy trials.

Objectives:

- To screen volunteers for clinical trials of vaccines or drugs to treat or prevent virus infections.

Eligibility:

- Healthy volunteers at least 18 years of age.

Design:

* Screening may begin several months before the start of the clinical trial. Participants may come to the National Institutes of Health clinic one or more times.
* Participants may be screened with a physical exam and medical history. Blood samples will be collected. Other samples may also be collected, including urine, nasal wash, nasal swab, or stool samples. All samples will be stored for reference by the study researchers....

DETAILED DESCRIPTION:
Vaccines and antiviral therapies are critical for prevention and treatment of viral diseases. Testing of vaccines, antiviral medications, or live virus challenge studies in volunteers may requires knowing whether the subject has been previously infected by the virus. We will recruit healthy persons for this study and screen them for their eligibility to participate in clinical trials of investigational vaccines or antiviral products, investigational studies of licensed products, or live virus challenge studies. In most cases this will involve a medical history, physical examination, and obtaining blood to test for antibodies to the virus being studied in a vaccine or antiviral therapy trial or live virus challenge study. In some cases blood may be tested for viral DNA or RNA and urine, stool, saliva, nasal swab, or nasopharyngeal wash secretions may be tested for viruses or antibodies to the virus. Additional testing, such as an electrocardiogram (EKG), chest radiograph (CXR), and pulmonary function tests (PFTs) may be done. Samples will also be stored for future research. This study should help us to identify a group of volunteers that will be eligible, based on testing for their prior exposure to viruses, to participate in vaccine or antiviral therapy trials, or live virus challenge studies, .conducted by the Laboratory of Infectious Diseases, NIAID at the NIH Clinical Center.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Age: 18 years of age or older
  2. Available to participate for the planned duration of the clinical trial for which the screening is being done
  3. Able and willing to complete the informed consent process
  4. Agree to participate in proceduresas needed for the clinical trial screening process.

EXCLUSION CRITERIA:

1. A known condition that requires active medical intervention or monitoring to avert serious danger to the participant s health or well-being
2. Known to be pregnant or breast-feeding, or planning to become pregnant in the near future
3. Use of a medication that significantly alters the immune system within the past 6 months or anticipated within the next year (e.g. immunoglobulin, systemic corticosteroids > prednisone equivalent of 10 mg/kg/day)
4. Any other condition that in the opinion of the investigator would make the subject unsuitable for enrollment or could interfere with the subject participating in and completing the study
5. Abuse of illicit drugs, alcohol abuse, or alcohol dependency within the last 6 months
6. Known to be infected with HIV or Hepatitis B and/or C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers aged 18 or older.
Sampling Method: Non-Probability Sample
Enrollment: 359 (Actual)
Dates: Start 2012-11-27 (Actual); Primary Completion 2021-07-21 (Actual); Study Completion 2021-07-21 (Actual)

PRIMARY OUTCOMES:
To screen subjects for their eligibility to participate in clinical trials of investigational or licensed vaccines, antiviral products, or live virus challenge studies being evaluated for research purposes. | At every patient contact.
  Eligibility will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey I Cohen, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2012-I-0121.html